CLINICAL TRIAL: NCT00816023
Title: CONSERV-1 (Clinical Outcomes and Safety Trial to Investigate Ecallantide's Effect on Reducing Surgical Blood Loss Volume) A Phase 2 Randomized Placebo-controlled Dose-ranging Study in Subjects Exposed to Cardio-pulmonary Bypass During Primary Coronary Artery Bypass Graft Surgery
Brief Title: A Dose-ranging Safety and Efficacy Study of Ecallantide to Reduce Surgical Blood Loss Volume
Acronym: CONSERV-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECAL-PCPB-08-02
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Bloodloss; Surgical Procedures, Operative
MeSH Terms: interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ecallantide Low Dose (Experimental): target steady state concentration of 0.15 mg/L
  Interventions: Drug: ecallantide
- Ecallantide Medium Dose (Experimental): target steady state concentration of 0.75 mg/L
  Interventions: Drug: ecallantide
- Ecallantide High Dose (Experimental): target steady state concentration of 2.25 mg/L
  Interventions: Drug: ecallantide
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ecallantide — infusion administered IV over the duration of the surgical procedure
  Arms: Ecallantide High Dose; Ecallantide Low Dose; Ecallantide Medium Dose
Drug: placebo — solution for IV infusion over the duration of the surgical>> procedure
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and identify the optimal dose(s) of ecallantide in reducing blood loss in subjects undergoing coronary artery bypass surgery including the use of cardio pulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (by study subject or appropriate legal representative) prior to any study-related procedure not part of normal medical care
* Planned primary CABG surgery including the use of cardio-pulmonary bypass.

Exclusion Criteria:

* Planned concomitant surgery including ASD repair, valve replacement, carotid endarterectomy, CABG combined procedures or any repeat sternotomy;
* Body weight <55 kg;
* Planned hypothermia (<28ºC);
* Planned transfusion in the peri-operative or post-operative periods;
* Planned transfusion of pre-operatively donated autologous blood;
* Female subjects who are pregnant or lactating;
* Planned use of desmopressin, lysine analogs, atrial natriuretic hormone or recombinant activated Factor VII;
* Planned use of corticosteroids in the pump prime solution;
* Ejection fraction <30% within 90 days prior to surgery;
* Evidence of a myocardial infarction within 5 days prior to surgery;
* History of stroke or transient ischemic attack within 3 months prior to surgery;
* Hypotension or heart failure requiring the use of inotropes or mechanical devices within 24 hours prior to surgery;
* Serum creatinine >2.0 mg/dL within 48 hours prior to surgery;
* Serum hepatic enzymes above 2.5 times the upper limit of normal for the applicable laboratory;
* Hematocrit <32% within 48 hours prior to surgery;
* Platelet count below the normal range for the applicable laboratory within 14 days prior to surgery;
* History of, or family history of, bleeding or clotting disorder or thrombophilia;
* History of heparin-induced thrombocytopenia;
* Prothrombin time and/or activated partial thromboplastin time >1.5 X normal range;
* Serious intercurrent illness or active infection;
* Any previous exposure to ecallantide;
* Receipt of an investigational drug or device 30 days prior to participation in the current study;
* Known allergy to any agent expected to be used in the intra-operative or post-operative periods; and
* Administration of: Eptifibatide within 6 hours prior to surgery, Tirofiban HCl within 6 hours prior to surgery, *Enoxaparin sodium or other low-molecular-weight heparin <24 hours prior to surgery, Clopidogrel within 5 days prior to surgery, Ticlopidine within 7 days prior to surgery, Abciximab within 5 days prior to surgery, *Bivalirudin, argatroban or lepirudin within 6 hours prior to surgery, *Fondaparinux within 72 hours prior to surgery, Prasugrel within 10 days prior to surgery [*Prophylactic use permitted for the prevention of deep vein thrombosis.]

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Wheeler, MD, MFPM, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (29):
- United States (21):
  - Cardio-Thoracic Surgeons PC, Birmingham, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - University of Colorado - Denver, Aurora, Colorado
  - Pepin Heart Hospital & Kiran Patel Research Institute, Tampa, Florida
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - MCVI - Covenant Medical Center, Saginaw, Michigan
  - MCVI - St. Mary's of Michigan, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's - Roosevelt Hospital Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - East Tennessee Cardiovascular Surgery Group, Knoxville, Tennessee
  - Texas Heart Institute, Houston, Texas
  - Sentara Heart Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Charleston Area Medical Center (CAMC), Charleston, West Virginia
- Canada (8):
  - Foothills Medical Centre, Calgary, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Hospital Laval), Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ecallantide Low Dose | Ecallantide Medium Dose | Ecallantide High Dose | Placebo
Started | 71 | 62 | 69 | 74
Completed Therapy | 65 | 59 | 61 | 63
Completed | 62 | 56 | 60 | 62
Not Completed | 9 | 6 | 9 | 12
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — assessments complete prior to window | 1 | 1 | 2 | 1
Not completed — Randomized Not Treated | 6 | 4 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecallantide Low Dose | Ecallantide Medium Dose | Ecallantide High Dose | Placebo | Total
Number analyzed (Participants) | 71 | 62 | 69 | 74 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.96) | 63.9 (9.40) | 63.2 (10.73) | 63.6 (10.90) | 63.4 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 15 | 11 | 54
  Male | 58 | 47 | 54 | 63 | 222
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 5 | 3 | 18
  White | 66 | 54 | 61 | 71 | 252
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Volume of Packed Red Blood Cells Transfused at 12 Hours Post Surgery
Time Frame: Start of surgery up to 12 hours after the end of surgery
Population: The Modified Intent to Treat population was the basis of this analysis, defined as all randomized subjects who received any amount of study drug and analyzed according to the planned treatment assignment.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ecallantide Low Dose | Ecallantide Medium Dose | Ecallantide High Dose | Placebo
Number analyzed (Participants) | 65 | 58 | 63 | 63
mL | 401.9 (624.87) | 383.1 (620.62) | 410.3 (639.47) | 377.6 (608.54)
Statistical Analysis 1: Comparison: Ecallantide Low Dose vs Ecallantide Medium Dose vs Ecallantide High Dose vs Placebo; Test type: Superiority or Other; p = 0.474, Jonckheere-Terpstra

2. Secondary Outcome: Treatment-emergent Adverse Events
Time Frame: Over the duration of the study.
Population: Analysis conducted on Safety population, defined as all subjects randomized and received any study drug. Treatment groups are based on actual treatment received.
Measure: Number; unit: participants
Arm/Group | Ecallantide Low Dose | Ecallantide Medium Dose | Ecallantide High Dose | Placebo
Number analyzed (Participants) | 65 | 59 | 62 | 63
participants
  At least 1 TEAE | 65 | 59 | 62 | 63
  At least 1 Treatment-related AE | 7 | 9 | 4 | 7
  At least 1 AE of Severe Intensity | 11 | 13 | 15 | 16
  At least 1 Treatment-emergent SAE | 15 | 19 | 19 | 15
  At least 1 Treatment-related SAE | 1 | 3 | 1 | 1
  TEAE Resulting on Discontinuation of Study Drug | 0 | 0 | 1 | 0
  TEAE Resulting in Death | 0 | 1 | 0 | 0
  Treatment-related TEAE Resulting in Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | ECALLANTIDE HIGH DOSE | ECALLANTIDE MEDIUM DOSE | ECALLANTIDE LOW DOSE | PLACEBO
Serious Adverse Events (participants affected / at risk) | 19/62 | 19/59 | 15/65 | 15/63
Other Adverse Events (participants affected / at risk) | 62/62 | 59/59 | 65/65 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECALLANTIDE HIGH DOSE (N=62) | ECALLANTIDE MEDIUM DOSE (N=59) | ECALLANTIDE LOW DOSE (N=65) | PLACEBO (N=63)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3) | 2 (2) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 (6) | 4 (4) | 6 (6) | 3 (3)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECALLANTIDE HIGH DOSE (N=62) | ECALLANTIDE MEDIUM DOSE (N=59) | ECALLANTIDE LOW DOSE (N=65) | PLACEBO (N=63)
Anaemia (Blood and lymphatic system disorders) | 21 (21) | 30 (31) | 25 (28) | 22 (23)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8) | 5 (5) | 4 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 6 (6) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 18 (20) | 23 (23) | 17 (17) | 12 (12)
Atrial flutter (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 7 (7) | 8 (8) | 9 (9) | 11 (11)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (5) | 7 (7) | 3 (3) | 5 (5)
Ventricular extrasystoles (Cardiac disorders) | 7 (8) | 5 (6) | 2 (2) | 4 (5)
Constipation (Gastrointestinal disorders) | 24 (24) | 24 (24) | 20 (20) | 17 (17)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 31 (31) | 22 (23) | 30 (30) | 29 (29)
Vomiting (Gastrointestinal disorders) | 8 (9) | 5 (5) | 5 (5) | 2 (2)
Asthenia (General disorders) | 1 (1) | 5 (5) | 3 (3) | 1 (1)
Chills (General disorders) | 6 (6) | 4 (4) | 4 (4) | 3 (3)
Generalised oedema (General disorders) | 22 (22) | 22 (23) | 17 (17) | 16 (17)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Oedema (General disorders) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 7 (7) | 6 (6) | 8 (8) | 8 (8)
Pain (General disorders) | 5 (6) | 3 (3) | 5 (7) | 1 (1)
Pyrexia (General disorders) | 7 (7) | 14 (14) | 9 (9) | 8 (8)
Anaemia postoperative (Injury, poisoning and procedural complications) | 8 (8) | 5 (5) | 5 (5) | 4 (4)
Incision site pain (Injury, poisoning and procedural complications) | 18 (20) | 18 (19) | 14 (17) | 19 (19)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 4 (4)
Post procedural discharge (Injury, poisoning and procedural complications) | 5 (6) | 2 (2) | 2 (2) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 7 (7)
Procedural nausea (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 42 (43) | 36 (36) | 44 (44) | 37 (37)
Blood calcium decreased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 3 (3) | 4 (4) | 7 (7) | 2 (2)
Breath sounds abnormal (Investigations) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Urine output decreased (Investigations) | 4 (4) | 8 (8) | 5 (5) | 5 (5)
White blood cell count increased (Investigations) | 5 (5) | 6 (6) | 3 (3) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 5 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 27 (28) | 24 (24) | 23 (23) | 28 (28)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 4 (4) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (9) | 6 (6) | 4 (4) | 5 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5) | 2 (2) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9) | 7 (7) | 12 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 5 (5) | 1 (1)
Agitation (Psychiatric disorders) | 5 (6) | 3 (3) | 5 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4) | 9 (9) | 7 (7)
Confusional state (Psychiatric disorders) | 6 (6) | 3 (3) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 9 (9) | 12 (12) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 30 (32) | 26 (27) | 23 (24) | 28 (28)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 7 (7) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 18 (21) | 13 (14) | 17 (18)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 3 (3) | 7 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 5 (5)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (12) | 8 (8) | 5 (5)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 5 (5) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (3)
Hypertension (Vascular disorders) | 8 (8) | 8 (8) | 10 (10) | 7 (7)
Hypotension (Vascular disorders) | 24 (25) | 25 (26) | 28 (31) | 17 (17)

LIMITATIONS AND CAVEATS:
Secondary efficacy variables were considered exploratory and, based on failure of the primary endpoint to meet statistical significance and early termination of the trial, are not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If the First Publication is not published within 1 year of Study conclusion or termination, Investigator shall have the right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.